CLINICAL TRIAL: NCT03182101
Title: Quality Assessment in Exposure Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bradley Hospital (Other)
Responsible Party: Principal Investigator, Kristen Benito, Principle Investigator, Bradley Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1039342
Record Dates: First submitted 2017-06-01; First posted 2017-06-09 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Obsessive-Compulsive Disorder in Children
MeSH Terms: interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure Therapy with fidelity checklist (Experimental): Therapist and parent/child participants will complete an Exposure Guide after each session.
  Interventions: Behavioral: Exposure Therapy

INTERVENTIONS:
Behavioral: Exposure Therapy — Exposure Therapy is a form of Cognitive Behavioral Therapy. There is strong evidence for exposure as a necessary and primary ingredient for treating anxiety and OCD, and exposure is the most common practice element in treatment protocols for anxiety.

SUMMARY:
This project will test a measure of treatment quality, Exposure Guide, for therapists using exposure therapy for youths and young adults with anxiety or OCD. We anticipate that users of this measure will be able to complete it reliably, find it acceptable, and that the measure will predict patient outcome. This project will include 40 therapists treating 300 anxious youth and young adults ages 5-25 at a large community mental health agency. Results of this study will establish the Exposure Guide as a measure of exposure quality in real world settings.

DETAILED DESCRIPTION:
Empirically supported behavioral treatments cannot be effectively disseminated without understanding key quality components. Mechanism-informed quality measures have extraordinary potential to enhance pragmatism by eliminating unnecessary elements and targeting multiple problems and populations, and to enhance predictive value by detecting mechanism engagement early in treatment. Community Mental Health Agencies (CMHAs), however, are often ill-equipped to use such measures of treatment quality due to burden and limited resources. Exposure therapy for anxiety is an ideal prototype for testing a practical, mechanism-informed quality measure in CMHAs given its potential for public health impact and clear theory of mechanism. The Exposure Guide (EG), a brief quality tool measuring therapist behaviors and mechanism, was developed based on microanalytic coded data showing a strong link between therapist behavior and patient outcome across three RCTs of exposure therapy in youth. Initial psychometrics for the EG using these RCT data are promising showing reliability, construct validity, and predictive validity, and pilot data suggests it may be acceptable and feasible in a community setting. Building upon these findings, we propose to test this novel measure of exposure quality, EG, in a community setting including its reliability and validity, its pragmatism, and which community end-users can become reliable and valid reporters. Therapists at a large local CMHA (N = 40) treating anxious youth and young adults ages 5-25 (N = 300) will participate in this study. The EG will be completed by 1) agency supervisors monthly, 2) therapists per session, 3) patient/families per session, and 4) study raters per session. Results from this study will establish an innovative model for measuring therapeutic elements that trigger mechanism of change in real-world therapy as well as inform future use of EG as a training tool to improve exposure quality in community settings.

ELIGIBILITY:
Inclusion Criteria:

* Patient at a Community Mental Health Agency that is partnering with this study
* Primary or co-primary diagnosis of OCD, Separation Anxiety, Social Anxiety, Panic Disorder, or Specific Phobia.
* Children < age 12 have a caretaker available to participate in treatment
* Patient and parent/legal guardian are English speaking

Exclusion Criteria:

* Concurrent psychotherapy for treatment of anxiety
* Psychosis, Pervasive Developmental Disorder, or Mental Retardation

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Scales | Through study completion, an average of 6 months
  The Clinical Global Impression Scales (CGI) are brief, clinician-rated measures of global severity and improvement in treatment for children and adults.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Benito, PhD, Principal Investigator — The Warren Alpert Medical School of Brown University
Locations (1):
- Emma Pendleton Bradley Hospital, Riverside, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Twice yearly data sharing through NDCT
Time Frame: Secondary outcome data will be uploaded biannually beginning in January of 2018. Primary outcomes will be made available within 6 months of study completion.